CLINICAL TRIAL: NCT02466620
Title: A Comparison of Paediatric Weight Estimation Methods for Emergency Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 719/2557(EC4)
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Body Weight
Keywords: Body Weight; Resuscitation; Pediatric weight estimation
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the validity, reliability and practicality of the different weight estimation methods (parent estimation method, Mercy method, Broselow tape, original and update APLS) in Thai children.

DETAILED DESCRIPTION:
A reliable paediatric weight estimation method is crucial for the physician attempting to resuscitate an injured child. When a patient is in a critical, life threatening condition or in mass casualty settings, actual body weight cannot be obtained by weight measurement instrument. Several resuscitation modalities, such as resuscitation medications, fluid replacement, and amount of electrical shock in defibrillation, are calculated according to patient body weight

Besides from weight derived from children's parent which cannot achieve in some situations and vary in accuracy, Broselow tape is the gold standard currently for appraise children's weight from their length. However, this tape tends to underestimate weight and it is limited to use in children are less than 146 centimeters in length. Age- based weight estimation methods are the mathematical formulas to estimate weight from the children's age. The various methods described in the Advanced Paediatric Life support (APLS) both original and updated still have doubts about the accuracy and reliability. Both length- based and aged- based methods fail to resolve the overweight or obese and underweight children who have the same height or the same age. Mercy method is the new weight estimation method that incorporates the humeral length and mid-upper arm circumference to estimate the child weight. This method has been demonstrated both accuracy and reliability over other existing methods. This study will evaluate the validity, reliability and practicality of the previously mentioned pediatric weight estimation methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Informed consent and assent (7-12 years) were obtained

Exclusion Criteria:

* Disabling children
* Incapable to stand up or lie down to measure weight or length
* Chronic steroid use
* Edema from known diseases
* Extremities joint contracture

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 2 sources of study population:
  1. Children from pre-school and primary school at Wat Amarintararam School, Bangkok, Thailand
  2. Children from the out-patient department at Siriraj hospital, Bangkok, Thailand
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The validity of the different weight estimation methods | at time of measurement within one day
  The performance of the Mercy method, Broselow tape, parental estimation and aged-base methods (original APLS,updated APLS formula) were compared against the actual weight and against each other. Agreement between estimated weight and actual weight of each weight estimation method was determined by Bland-Altman plots with 95% limits of agreement and correlation test. Bias and variability tested by calculate error : predicted weight -actual weight, calculated percentage error : [(predicted - actual weight) x 100%] / actual weight, calculated root mean square error = square root of the average squared error. Categorical error analysis was done by the percentage error of each of the estimation techniques within 10% and 20% of actual weight.

SECONDARY OUTCOMES:
The reliability of the different weight estimation methods | at time of measurement within one day
  The inter-rater reliability compared the results between two raters. The intra-rater reliability was compared the results from first and second measurement in one rater.The value was tested by intra- class correlation coefficient that a value > 0.8 was considered to excellent correlation.
The practicality of the different weight estimation methods | at time of measurement within one day
  User satisfaction was evaluated from questionnaire and the values were analysed by descriptive statistics. Time from start measurement until get the estimated weight was recorded in all methods (except in parental estimation method) to calculate median time measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Artid Samerchua, Principal Investigator — Mahidol University
Locations (1):
- Artid Samerchua, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Lundahl A, Kidwell KM, Nelson TD. Parental underestimates of child weight: a meta-analysis. Pediatrics. 2014 Mar;133(3):e689-703. doi: 10.1542/peds.2013-2690. Epub 2014 Feb 2. PMID 24488736
- [Background] Graves L, Chayen G, Peat J, O'Leary F. A comparison of actual to estimated weights in Australian children attending a tertiary children's' hospital, using the original and updated APLS, Luscombe and Owens, Best Guess formulae and the Broselow tape. Resuscitation. 2014 Mar;85(3):392-6. doi: 10.1016/j.resuscitation.2013.11.024. Epub 2013 Dec 7. PMID 24321321
- [Background] Dicko A, Alhousseini ML, Sidibe B, Traore M, Abdel-Rahman SM. Evaluation of the Mercy weight estimation method in Ouelessebougou, Mali. BMC Public Health. 2014 Mar 21;14:270. doi: 10.1186/1471-2458-14-270. PMID 24650051
- [Background] Abdel-Rahman SM, Ridge A, Kearns GL. Estimation of body weight in children in the absence of scales: a necessary measurement to insure accurate drug dosing. Arch Dis Child. 2014 Jun;99(6):570-4. doi: 10.1136/archdischild-2013-305211. Epub 2014 Feb 26. No abstract available. PMID 24573883
- [Background] Abdel-Rahman SM, Ahlers N, Holmes A, Wright K, Harris A, Weigel J, Hill T, Baird K, Michaels M, Kearns GL. Validation of an improved pediatric weight estimation strategy. J Pediatr Pharmacol Ther. 2013 Apr;18(2):112-21. doi: 10.5863/1551-6776-18.2.112. PMID 23798905
- [Background] Trakulsrichai S, Boonsri C, Chatchaipun P, Chunharas A. Accuracy of three methods used for Thai children's body weight estimation. J Med Assoc Thai. 2012 Sep;95(9):1194-9. PMID 23140037
- [Background] Loo PY, Chong SL, Lek N, Bautista D, Ng KC. Evaluation of three paediatric weight estimation methods in Singapore. J Paediatr Child Health. 2013 Apr;49(4):E311-6. doi: 10.1111/jpc.12141. Epub 2013 Mar 14. PMID 23489439
- [Background] Meguerdichian MJ, Clapper TC. The Broselow tape as an effective medication dosing instrument: a review of the literature. J Pediatr Nurs. 2012 Aug;27(4):416-20. doi: 10.1016/j.pedn.2012.04.009. Epub 2012 May 8. No abstract available. PMID 22579781